CLINICAL TRIAL: NCT02470091
Title: Phase 2 Study of Denosumab (NSC# 744010), a RANK Ligand Antibody, for Recurrent or Refractory Osteosarcoma
Brief Title: Denosumab in Treating Patients With Recurrent or Refractory Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOST1321; NCI-2015-00543 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s15-01360; AOST1321; AOST1321 (Other: Children's Oncology Group); AOST1321 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-04-14; First posted 2015-06-12 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Osteosarcoma; Recurrent Osteosarcoma; Refractory Osteosarcoma; Stage IV Osteosarcoma AJCC v7; Stage IVA Osteosarcoma AJCC v7; Stage IVB Osteosarcoma AJCC v7
MeSH Terms: conditions — Osteosarcoma | interventions — Denosumab; QL1206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (denosumab) (Experimental): Patients receive denosumab SC on day 1 (days 1, 8, and 15 of course 1 only). Treatment repeats every 4 weeks (28 days) for up to 24 months or 26 courses, whichever occurs first, in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Denosumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Denosumab — Given SC
  Other Names: AMG 162; AMG-162; Denosumab Biosimilar MW032; Denosumab Biosimilar QL1206; Denosumab Biosimilar TK-006; Prolia; TK-006; Xgeva
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well denosumab works in treating patients with osteosarcoma that has come back (recurrent) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as denosumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether denosumab therapy either increases the disease control rate at 4 months in patients with recurrent measurable osteosarcoma as compared to historical Children's Oncology Group (COG) experience or denosumab therapy produces an objective response rate greater than 5% (Cohort 1).

II. To determine whether denosumab therapy increases the disease control rate at 12 months in patients with recurrent resected osteosarcoma as compared to historical COG experience (Cohort 2).

SECONDARY OBJECTIVES:

I. To investigate the pharmacokinetics (PK) and pharmacodynamics (PD) of denosumab in subjects with recurrent osteosarcoma.

II. To describe the tolerability of denosumab in subjects with recurrent osteosarcoma.

III. To report the disease control rate and objective response rate for patients with recurrent osteosarcoma limited to bone.

IV. To investigate biological markers potentially associated with response to denosumab in patients with recurrent osteosarcoma.

OUTLINE:

Patients receive denosumab subcutaneously (SC) on day 1 (days 1, 8, and 15 of course 1 only). Treatment repeats every 4 weeks (28 days) for up to 24 months or 26 courses, whichever occurs first, in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Female patients must have a bone age of equal to or greater than 12 years of age as determined by local read of appropriate radiographic imaging
* Male patients must have a bone age of equal to or greater than 14 years of age as determined by local read of appropriate radiographic imaging
* Patients must have relapsed or become refractory to conventional therapy, with a regimen including some combination of high dose methotrexate, doxorubicin, cisplatin, ifosfamide and etoposide; and have had histologic verification of osteosarcoma at original diagnosis or at the time of recurrence
* Cohort 1 patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Cohort 2 patients must have had a complete resection of all sites of metastatic disease within 30 days prior to enrollment

  * Patients will only be eligible after they have undergone complete surgical resection of suspected metastatic disease that is histopathologically confirmed to be osteosarcoma prior to enrollment

    * Note: the definition of complete resections is: gross resection of all disease as per the operating surgeon; post-operative imaging is not required for confirmation of complete resection
  * Patients must undergo resection of any lung lesion meeting criteria for likely metastatic disease, defined as:

    * 3 or more lesions > 5 mm in diameter OR a single lesion > 1 cm
  * Patients with lung as the only site of resected metastatic disease must have refused participation in protocol AOST1421

    * Note: This applies if AOST1421 is open to enrollment at the enrolling institution on the day the patient consents
* Patient must have adequate tumor specimen available for submission
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: 11 to < 13 years old; 1.2 (male, female) maximum serum creatinine (mg/dL)
  * Age: 13 to < 16 years old; 1.5 (male), 1.4 (female) maximum serum creatinine (mg/dL)
  * Age: >= 16 years old; 1.7 (male), 1.4 (female) maximum serum creatinine (mg/dL)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x ULN for age
* Serum calcium or albumin-adjusted serum calcium >= 2.0 mmol/L (8.0 mg/dL) and =< 2.9 mmol/L (11.5 mg/dL)

Exclusion Criteria:

* Patients with known sensitivity to any of the products to be administered during the study (eg, mammalian derived products, calcium or vitamin D)
* Patients who are receiving other cancer directed therapy at the time of enrollment
* Patients who have previously received denosumab
* Patients who have previously received mithramycin, strontium-89, samarium-153 or rhenium
* Patients receiving bisphosphonates
* Pre-existing conditions

  * Disorders associated with abnormal bone metabolism
  * Hypocalcemia that is not corrected with oral calcium supplementation
  * Vitamin D < 20 mg/mL
  * Paget's disease
  * Prior history or current evidence of osteonecrosis of the jaw
  * Any dental or oral condition likely to result in disruption of mucosal integrity during denosumab therapy including: active dental or jaw condition requiring oral surgery or tooth extraction; non-healed dental or oral surgery or planned invasive dental procedures during the anticipated course of study therapy
  * Unstable systemic disease, excluding osteosarcoma, such as unstable proximal renal tubule dysfunction (Fanconi syndrome) or congestive heart failure
* Pregnancy and breast feeding

  * Female patients who are pregnant; a pregnancy test is required for female patients of childbearing potential
  * Lactating females who plan to breastfeed their infants while on study therapy and through 5 months after completion of study therapy
  * Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 5 months after the end of study treatment
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 11 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Janeway, Principal Investigator — Children's Oncology Group
Locations (141):
- United States (132):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Centralia Oncology Clinic, Centralia, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Measurable: Cohort 1 patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
- Cohort 2: Resection: Cohort 2 patients must have had a complete resection of all sites of metastatic disease within 30 days prior to enrollment
Period: Overall Study
Arm/Group | Cohort 1: Measurable | Cohort 2: Resection
Started | 16 | 40
Follow-up Report | 1 | 10
Completed | 15 | 38
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Measurable | Cohort 2: Resection | Total
Number analyzed (Participants) | 16 | 40 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 26 | 42
  Between 18 and 65 years | 0 | 14 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 15 [11 to 17] | 17 [12 to 36] | 16 [11 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 17 | 22
  Male | 11 | 23 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 10 | 32 | 42
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 32 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 16 | 39 | 55
  Canada | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (Cohort I)
Description: Disease control interval was calculated as the time from enrolment until detection of new disease or progression of an existing site of disease as determined by the treating physician. Disease control interval of at least 4 months was considered disease control success.
Time Frame: At 4 months
Population: 1 patient was excluded due to withdrawal.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Measurable
Number analyzed (Participants) | 15
participants | 1

2. Primary Outcome: Response Evaluation Criteria in Solid Tumors (RECIST) Response (Complete Response [CR] or Partial Response [PR] vs Not CR or PR) (Cohort I)
Description: Per Response Evaluation Criteria In Solid TumorsCriteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response(CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At 4 months
Population: 1 patient was excluded due to withdrawal.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Measurable
Number analyzed (Participants) | 15
participants | 0

3. Primary Outcome: Disease Control Rate (Cohort II)
Description: Disease control interval was calculated as the time from enrolment until detection of new disease as determined by the treating physician. Disease control interval of at least 12 months was considered disease control success.
Time Frame: At 12 months
Population: 2 patients were excluded due to ineligibility
Measure: Number; unit: participants
Arm/Group | Cohort 2: Resection
Number analyzed (Participants) | 38
participants | 10

4. Secondary Outcome: Pharmacokinetic (PK) Parameters: Mean of Trough Concentrations of Denosumab
Description: Sample means of trough concentrations of denosumab will be calculated.
Time Frame: Days 1, 8, 15, and 22 of course 1, day 1 of courses 2-4 and 7, and days 1 and 15 of course 6
Population: The number of patients who contributed samples varied across cycles.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1: Measurable | Cohort 2: Resection
Number analyzed (Participants) | 15 | 27
ng/ml
  Serum denosumab (ng/ml): Cycle 1, Day 1 | 0 (0) | 0 (0)
  Serum denosumab (ng/ml): Cycle 1, Day 8: number analyzed (Participants) | 13 | 26
  Serum denosumab (ng/ml): Cycle 1, Day 8 | 11.59 (3.836665219) | 10.81 (4.514421336)
  Serum denosumab (ng/ml): Cycle 1, Day 15: number analyzed (Participants) | 12 | 24
  Serum denosumab (ng/ml): Cycle 1, Day 15 | 20.57 (8.290958931) | 22.07 (10.0339424)
  Serum denosumab (ng/ml): Cycle 1, Day 22: number analyzed (Participants) | 10 | 25
  Serum denosumab (ng/ml): Cycle 1, Day 22 | 31.8 (12.85573802) | 31.56 (13.41044369)
  Serum denosumab (ng/ml): Cycle 2, Day 1: number analyzed (Participants) | 10 | 24
  Serum denosumab (ng/ml): Cycle 2, Day 1 | 30.57 (10.78239306) | 30.28 (11.77497346)
  Serum denosumab (ng/ml): Cycle 3, Day 1: number analyzed (Participants) | 1 | 16
  Serum denosumab (ng/ml): Cycle 3, Day 1 | 23.8 (NA) — Only 1 participant was analyzed | 27.49 (13.31277582)
  Serum denosumab (ng/ml): Cycle 4, Day 1: number analyzed (Participants) | 1 | 14
  Serum denosumab (ng/ml): Cycle 4, Day 1 | 23.7 (NA) — Only 1 participant was analyzed | 23.67 (11.83849653)
  Serum denosumab (ng/ml): Cycle 6, Day 1: number analyzed (Participants) | 1 | 6
  Serum denosumab (ng/ml): Cycle 6, Day 1 | 20.3 (NA) — Only 1 participant was analyzed | 31.22 (14.57292009)
  Serum denosumab (ng/ml): Cycle 6, Day 15: number analyzed (Participants) | 1 | 10
  Serum denosumab (ng/ml): Cycle 6, Day 15 | 23.2 (NA) — Only 1 participant was analyzed | 26.66 (11.95742447)
  Serum denosumab (ng/ml): Cycle 7, Day 1: number analyzed (Participants) | 0 | 6
  Serum denosumab (ng/ml): Cycle 7, Day 1 |  | 30.22 (13.89748179)

5. Secondary Outcome: Pharmacokinetic (PK) Parameters: Median of Trough Concentrations of Denosumab
Description: Sample medians of trough concentrations of denosumab will be calculated.
Time Frame: Days 1, 8, 15, and 22 of course 1, day 1 of courses 2-4 and 7, and days 1 and 15 of course 6
Population: The number of patients who contributed samples varied across cycles.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Cohort 1: Measurable | Cohort 2: Resection
Number analyzed (Participants) | 15 | 27
ng/ml
  Serum denosumab (ng/ml): Cycle 1, Day 1 | 0 [0 to 0] | 0 [0 to 0]
  Serum denosumab (ng/ml): Cycle 1, Day 8: number analyzed (Participants) | 13 | 26
  Serum denosumab (ng/ml): Cycle 1, Day 8 | 10.8 [5.54 to 19.8] | 9.34 [6.23 to 25.1]
  Serum denosumab (ng/ml): Cycle 1, Day 15: number analyzed (Participants) | 12 | 24
  Serum denosumab (ng/ml): Cycle 1, Day 15 | 20.7 [5.96 to 35.7] | 18.75 [12.9 to 54.5]
  Serum denosumab (ng/ml): Cycle 1, Day 22: number analyzed (Participants) | 10 | 25
  Serum denosumab (ng/ml): Cycle 1, Day 22 | 27.85 [15.2 to 57.6] | 27.6 [17.1 to 74]
  Serum denosumab (ng/ml): Cycle 2, Day 1: number analyzed (Participants) | 10 | 24
  Serum denosumab (ng/ml): Cycle 2, Day 1 | 30.75 [13.6 to 49.9] | 27.3 [17 to 63.3]
  Serum denosumab (ng/ml): Cycle 3, Day 1: number analyzed (Participants) | 1 | 16
  Serum denosumab (ng/ml): Cycle 3, Day 1 | 23.8 [23.8 to 23.8] | 22.8 [13.8 to 61]
  Serum denosumab (ng/ml): Cycle 4, Day 1: number analyzed (Participants) | 1 | 14
  Serum denosumab (ng/ml): Cycle 4, Day 1 | 23.7 [23.7 to 23.7] | 21.6 [10.6 to 48.8]
  Serum denosumab (ng/ml): Cycle 6, Day 1: number analyzed (Participants) | 1 | 6
  Serum denosumab (ng/ml): Cycle 6, Day 1 | 20.3 [20.3 to 20.3] | 32.05 [14.9 to 51.5]
  Serum denosumab (ng/ml): Cycle 6, Day 15: number analyzed (Participants) | 1 | 10
  Serum denosumab (ng/ml): Cycle 6, Day 15 | 23.2 [23.2 to 23.2] | 23.5 [12.1 to 49.1]
  Serum denosumab (ng/ml): Cycle 7, Day 1: number analyzed (Participants) | 0 | 6
  Serum denosumab (ng/ml): Cycle 7, Day 1 |  | 27.95 [17.9 to 56.5]

6. Secondary Outcome: Pharmacodynamic (PD) Parameters of Denosumab: Serum C-telopeptide
Description: Serum c-telopeptide in pg/ml
Time Frame: Days 1, 8, 15, and 22 of course 1 and day 1 of courses 2-4 and 7
Population: All eligible participants
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Cohort 1: Measurable | Cohort 2: Resection
Number analyzed (Participants) | 15 | 38
pg/ml
  Serum c-telopeptide (pg/ml): Cycle 1, Day 1: number analyzed (Participants) | 15 | 34
  Serum c-telopeptide (pg/ml): Cycle 1, Day 1 | 1713 (1857) | 944.5 (543)
  Serum c-telopeptide (pg/ml): Cycle 1, Day 8: number analyzed (Participants) | 12 | 32
  Serum c-telopeptide (pg/ml): Cycle 1, Day 8 | 220.5 (77) | 244.0625 (259)
  Serum c-telopeptide (pg/ml): Cycle 1, Day 15: number analyzed (Participants) | 11 | 15
  Serum c-telopeptide (pg/ml): Cycle 1, Day 15 | 203.1818 (68) | 171.24 (86)
  Serum c-telopeptide (pg/ml): Cycle 1, Day 22: number analyzed (Participants) | 9 | 30
  Serum c-telopeptide (pg/ml): Cycle 1, Day 22 | 210.8889 (95) | 178.5033 (96)
  Serum c-telopeptide (pg/ml): Cycle 2, Day 1: number analyzed (Participants) | 10 | 31
  Serum c-telopeptide (pg/ml): Cycle 2, Day 1 | 200.8 (78) | 152.2032 (61)
  Serum c-telopeptide (pg/ml): Cycle 3, Day 1: number analyzed (Participants) | 1 | 22
  Serum c-telopeptide (pg/ml): Cycle 3, Day 1 | 115 | 147.8818 (85)
  Serum c-telopeptide (pg/ml): Cycle 4, Day 1: number analyzed (Participants) | 1 | 17
  Serum c-telopeptide (pg/ml): Cycle 4, Day 1 | 116 | 137.0235 (80)
  Serum c-telopeptide (pg/ml): Cycle 7, Day 1: number analyzed (Participants) | 1 | 10
  Serum c-telopeptide (pg/ml): Cycle 7, Day 1 | 108 | 168.9 (81)

7. Secondary Outcome: Pharmacodynamic (PD) Parameters of Denosumab: Urine N-telopeptide to Creatinine Ratio
Description: Urine n-telopeptide to creatinine ratio expressed as nMol BCE/mmol creatinine
Time Frame: Days 1, 8, 15, and 22 of course 1 and day 1 of courses 2-4 and 7
Population: All eligible participants
Measure: Mean (Standard Deviation); unit: nMol BCE/mmol creatinine
Arm/Group | Cohort 1: Measurable | Cohort 2: Resection
Number analyzed (Participants) | 15 | 38
nMol BCE/mmol creatinine
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 1: number analyzed (Participants) | 15 | 35
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 1 | 322.2 (307) | 190.7714 (283)
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 8: number analyzed (Participants) | 11 | 32
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 8 | 30.36364 (20) | 34.1875 (35)
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 15: number analyzed (Participants) | 11 | 30
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 15 | 26.18182 (14) | 32.3 (36)
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 22: number analyzed (Participants) | 9 | 31
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 1, Day 22 | 26.55556 (19) | 32.16129 (40)
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 2, Day 1: number analyzed (Participants) | 10 | 28
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 2, Day 1 | 22.1 (15) | 28.42857 (45)
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 3, Day 1: number analyzed (Participants) | 1 | 21
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 3, Day 1 | 14 | 24.7619 (20)
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 4, Day 1: number analyzed (Participants) | 1 | 17
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 4, Day 1 | 20 | 29.29412 (31)
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 7, Day 1: number analyzed (Participants) | 1 | 10
  Urine n-telopeptide to creatinine ratio (nMol BCE/mmol creatinine): Cycle 7, Day 1 | 13 | 22.4 (18)

8. Secondary Outcome: Incidence of Adverse Events, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The number of cycles where a dose-limiting toxicity was identified where dose-limiting toxicity is defined in the protocol using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Minimum of 2 years
Population: 56 patients were treated on protocol therapy. Three hundred seventy-three cycles were reported for the analysis of dose limiting toxicity
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | Treatment (Denosumab)
Number analyzed (Participants) | 56
Number analyzed (cycles) | 373
cycles | 1

9. Secondary Outcome: Response Rate (CR or PR) for Patients With Recurrent Osteosarcoma Limited to Bone (Cohort I)
Description: Confidence intervals will be constructed using the approximate normal distribution of each of the estimates and their asymptotic variances.
Time Frame: Up to 3 years post-treatment
Population: There were not any patients that met criteria for bone site
Arm/Group | Cohort 1: Measurable
Number analyzed (Participants) | 0

10. Secondary Outcome: Disease Control Rates for Patients With Recurrent Osteosarcoma Limited to Bone (Cohort I)
Description: as for outcome 9
Time Frame: At 4 months
Population: There were not any patients that met criteria for bone site
Arm/Group | Cohort 1: Measurable
Number analyzed (Participants) | 0

11. Secondary Outcome: Disease Control Rates for Patients With Recurrent Osteosarcoma Limited to Bone (Cohort II)
Description: Disease control interval was calculated at the time from enrolment until detection of new disease as determined by the treating physician. The proportion of patients who experience disease control of at least 12 months will be estimated by the method of Kaplan and Meier.
Time Frame: At 12 months
Population: Patients that met criteria for bone site
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Cohort 2: Resection
Number analyzed (Participants) | 6
proportion of patients | 0.667 [0.195 to 0.904]

ADVERSE EVENTS:
Time Frame: Through completion protocol therapy planned as 728 days after study enrollment
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Cohort 1: Measurable | Cohort 2: Resection
All-Cause Mortality (participants affected / at risk) | 13/15 | 20/38
Serious Adverse Events (participants affected / at risk) | 6/15 | 4/38
Other Adverse Events (participants affected / at risk) | 1/15 | 8/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Measurable (N=15) | Cohort 2: Resection (N=38)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Measurable (N=15) | Cohort 2: Resection (N=38)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT02470091/Prot_SAP_000.pdf